CLINICAL TRIAL: NCT06071611
Title: Cognitive Frailty and Oxygen-ozone Therapy: Integrated Approach to Identify Biological and Neuropsychological Markers
Brief Title: Cognitive Frailty and Oxygen-ozone Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Cristian Bonvicini, Co-Principal Investigator (CoPI), IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RF-2016-02363298
Record Dates: First submitted 2023-09-11; First posted 2023-10-06 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Frailty
MeSH Terms: interventions — Air

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxygen-Ozone (O2-O3) (Experimental): A small catheter is inserted into the rectum and a total amount of 150cc of O2-O3 mixture at the concentration of 30ug of O3 per cc of O2 over a 5-10 min period is administered.
  Interventions: Other: Experimental: Oxygen-Ozone (O2-O3)
- Oxygen (O2) (Active Comparator): A small catheter is inserted into the rectum and a total amount of 150cc of O2 over a 5-10 min period is administered.
  Interventions: Other: Active Comparator: Oxygen (O2)
- Placebo (Air) (Placebo Comparator): A small catheter is inserted into the rectum and a total amount of 150cc of air over a 5-10 min period is administered.
  Interventions: Other: Placebo Comparator: Placebo (Air)

INTERVENTIONS:
Other: Experimental: Oxygen-Ozone (O2-O3) — Oxygen-Ozone (O2-O3) treatment by rectal insufflations for 5 weeks (3 sessions for week).
  Arms: Oxygen-Ozone (O2-O3)
Other: Active Comparator: Oxygen (O2) — Oxygen (O2) treatment by rectal insufflations for 5 weeks (3 sessions for week).
  Arms: Oxygen (O2)
Other: Placebo Comparator: Placebo (Air) — Air treatment by rectal insufflations for 5 weeks (3 sessions for week).
  Arms: Placebo (Air)

SUMMARY:
As the world's population age, frailty is moving to the forefront of health and medical research and may become one of the world's most serious health issues. Understanding frailty prevention and treatment becomes even more crucial in order to reduce national healthcare costs. Oxygen-Ozone (O2-O3) therapy is a no-invasive/no-pharmacological and low cost procedure based on the therapeutic effects of low O3 concentrations, already used in medicine as an alternative/adjuvant treatment for different diseases and in the elderly. This project is the first pilot double blind randomized controlled trial where a group of elderly frail subjects are stratified as untreated (air), treated with pure O2 and treated with a mixture of O2-O3. The biological corollary will be transcriptomics, proteomics and also cognitive impairment assessment at baseline and after treatment. An algorithm combining these data will identify biomarkers of the response to O2-O3 therapy.

DETAILED DESCRIPTION:
Background: Although frailty does not yet have an internationally recognized standard definition, the general premise is that it may be considered a geriatric syndrome reflecting multi-system dysfunction, in which individuals are able to dynamically transition between severity states. The World Health Organization and The International Association of Geriatrics and Gerontology are working on an internationally accepted frailty definition. Accumulating evidence supports the existence of a close relation between frailty and cognitive impairment in subjects with/without dementia. To date specific treatments for the cognitive frailty are not still available. Oxygen-Ozone (O2-O3) therapy is a no-invasive/no-pharmacological low cost procedure based on therapeutic effects of low O3 concentrations and used in medicine as an alternative/adjuvant treatment for different diseases and for improving metabolic activities in elderly. Molecular evidence shows that low O3 concentrations dissolve in the biological fluids and induce a mild oxidative stress, which stimulates antioxidant defences thus preventing the inflammatory response and cell damage. Inflammatory processes, altered release of the main reactive O2 species and mitochondrial/cytoskeletal modifications have been hypothesized to influence significantly the frailty state as well as the neurodevelopmental network on cognitive impairment.

Aims

1. To characterize clinical and neuropsychological-cognitive impairment profiles in elderly frail subjects at baseline and after treatment.
2. To identify in vivo peripheral biomarkers associated to O2-O3 therapy through transcriptomic and proteomic analyses at baseline and after treatment.
3. To correlate clinical/cognitive improvement with transcriptomic and proteomic profiles to identify biomarkers associated to treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. subjects between the ages of 60 and 85, referring to the diagnosis of amnesic or non-amnesic cognitive disorder, reported by the subject himself or by family members;
2. MMSE score > 24/30;
3. exclusion of dementia, even in the presence of ascertained Alzheimer's disease detected by the most advanced diagnostic techniques;
4. function intact, or functional reduction not related to the cognitive problem;
5. pharmacological therapy for the treatment of stable cognitive or behavioral disorders for at least 3 months at the time of enrolment;
6. specific assessments/tools for frailty: "Italian frailty index (IFi)" and for "Frailty Instrument (FIt) based on the Survey of Health, Ageing and Retirement in Europe (SHARE-FIt)".

Exclusion Criteria:

1. subjects affected by disabling vision or hearing impairments;
2. subjects affected by known psychosis or psychiatric illness, alcohol or drug abuse;
3. subjects affected by uncontrolled hyperthyroidism or by Glucose-6-Phostate Dehydrogenase Deficiency (G6PD)-Favism (according to S.I.O.O.T Guidelines, http://www.ossiozono.it);
4. subjects who considered invasive the methodology for rectal insufflation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline and post-intervention in Italian frailty index (IFi) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Italian frailty index (IFi) is an Italian version of the "frailty index" based on accumulation of age-related deficits. IFi has been expressed as a ratio of deficits present/deficits considered after a comprehensive geriatric assessment.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Frailty Instrument (FIt) based on the Survey of Health, Ageing and Retirement in Europe (SHARE-FIt) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  SHARE-FIt is based on 5-item (i.e. grip strength and four self-reported items: fatigue, loss of appetite and/or eating less than usual, difficulties climbing stairs and/or walking 100 metres, and low level of physical activity). For each gender, a discreet factor (DFactor) model was estimated based on the five SHARE frailty variables.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Everyday Memory Questionnaire (EMQ) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Everyday Memory Questionnaire (EMQ) is a subjective measure of memory failure in everyday life, lower scores indicating better memory function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Raven's Progressive Matrices (RPM) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Raven's Progressive Matrices (RPM) is used to measure fluid intelligence, with higher scores indicating better function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Free and Cued Selective Reminding Test (FCSRT) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Free and Cued Selective Reminding Test (FCSRT) is a test used to assess episodic memory, with higher scores indicating better function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Rey-Osterrieth Complex Figure A Test (ROCF-A) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  ROCF-A is used to explore visuo-constructional ability and visuo-spatial memory, with higher scores indicating better function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Face-name association task (FNAT) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  FNAT is used to assess the patient's associative memory and is composed of encoding and retrieval phases, with higher scores indicating better function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Picture naming task (PNT) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  The PNT is designed to explore lexical access, with higher scores indicating better function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Trail Making Tests A (TMT-A) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Trail Making Tests A (TMT-A) is used to assess visual attention and motor speed skills, with lower scores indicating better attention.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in Trail Making Tests B (TMT-B) | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Trail Making Tests B (TMT-B) is used to assess executive functions, with lower scores indicating good performance in executive function.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score

SECONDARY OUTCOMES:
Change from baseline and post-intervention in peripheral mRNAs levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  The mRNAs peripheral signatures compared before and after treatments. To identify the list of differentially expressed mRNAs we filter ANOVA results using both fold change |FC| ≥ 1.5 and p-value ≤0.05.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral NGFb (beta-Nerve Growth Factor) levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of NGFb compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral BDNF (Brain Derived Neurotrophic Factor) levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of BDNF compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral VEGF (Vascular Endothelial Growth Factor) levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of VEGF compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-1b levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-1b compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-4 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-4 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-6 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-6 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-8 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-8 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-9 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-9 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-10 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-10 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IL, Interleukin-13 levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IL-13 compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral TNF-a (Tumor Necrosis Factor) levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of TNF-a compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score
Change from baseline and post-intervention in peripheral IFN-g (Interferon-gamma) levels in subjects stratified according to IFi or SHARE-FIt scores | Baseline (pre-intervention), post-intervention (3, 9 and 15 months)
  Peripheral concentrations (pg/ml) of IFN-g compared before and after treatments.
  Change = month 3rd after treatment - baseline score / Change = month 9th after treatment - baseline score / Change = month 15th after treatment - baseline score

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Geroldi, MD, Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (1):
- IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scassellati C, Ciani M, Galoforo AC, Zanardini R, Bonvicini C, Geroldi C. Molecular mechanisms in cognitive frailty: potential therapeutic targets for oxygen-ozone treatment. Mech Ageing Dev. 2020 Mar;186:111210. doi: 10.1016/j.mad.2020.111210. Epub 2020 Jan 23. PMID 31982474
- [Background] Scassellati C, Galoforo AC, Bonvicini C, Esposito C, Ricevuti G. Ozone: a natural bioactive molecule with antioxidant property as potential new strategy in aging and in neurodegenerative disorders. Ageing Res Rev. 2020 Nov;63:101138. doi: 10.1016/j.arr.2020.101138. Epub 2020 Aug 15. PMID 32810649
- [Background] Scassellati C, Galoforo AC, Esposito C, Ciani M, Ricevuti G, Bonvicini C. Promising Intervention Approaches to Potentially Resolve Neuroinflammation And Steroid Hormones Alterations in Alzheimer's Disease and Its Neuropsychiatric Symptoms. Aging Dis. 2021 Aug 1;12(5):1337-1357. doi: 10.14336/AD.2021.0122. eCollection 2021 Aug. PMID 34341712
- [Background] Varesi A, Chirumbolo S, Campagnoli LIM, Pierella E, Piccini GB, Carrara A, Ricevuti G, Scassellati C, Bonvicini C, Pascale A. The Role of Antioxidants in the Interplay between Oxidative Stress and Senescence. Antioxidants (Basel). 2022 Jun 22;11(7):1224. doi: 10.3390/antiox11071224. PMID 35883714
- [Background] Scassellati C, Costanzo M, Cisterna B, Nodari A, Galie M, Cattaneo A, Covi V, Tabaracci G, Bonvicini C, Malatesta M. Effects of mild ozonisation on gene expression and nuclear domains organization in vitro. Toxicol In Vitro. 2017 Oct;44:100-110. doi: 10.1016/j.tiv.2017.06.021. Epub 2017 Jun 23. PMID 28652203